CLINICAL TRIAL: NCT01393444
Title: Acute Electrocorticography (ECoG) Direct Brain Interface for Individuals With Upper Limb Paralysis
Brief Title: ECoG Direct Brain Interface for Individuals With Upper Limb Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer Collinger, PhD, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PRO10010149
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Tetraplegia; Spinal Cord Injury; Brachial Plexus Injury; Muscular Dystrophy; ALS; Brainstem Stroke
Keywords: Electrocorticography; Tetraplegia; Spinal cord injury; Brainstem stroke; Neuroprosthetic; Brain-computer interface; Direct brain interface; Neural activity; Motor cortex
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries; Muscular Dystrophies; Brain Stem Infarctions | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Direct Brain Interface Users (Experimental): All participants enrolled in the study will undergo "Implantation of ECoG sensors on the brain surface" to record neural activity. There is no control group. There are no other arms.
  Interventions: Device: Implantation of ECoG sensors on the brain surface

INTERVENTIONS:
Device: Implantation of ECoG sensors on the brain surface — One ECoG sensor will be implanted over the motor cortex of study participants
  Other Names: brain-computer interface; neuroprosthetic

SUMMARY:
The purpose of this research study is to demonstrate that individuals with upper limb paralysis due to spinal cord injury, brachial plexus injury, amyotrophic lateral sclerosis and brain stem stroke can successfully achieve direct brain control of assistive devices using an electrocorticography (ECoG)-based brain computer interface system.

DETAILED DESCRIPTION:
Brain-computer interface (BCI) technology aims to establish a direct link for transmitting information between the brain and external devices, offering a natural and rich control signal for prosthetic hands or functional electrical stimulators (FES) to re-animate paralyzed hands. This study focuses on an ECoG-based BCI system. ECoG measures brain activity using electrodes implanted on the surface of the brain. Each participant will undergo testing of the ECoG direct brain interface for up to 29 days. Participants will learn to control computer cursors, virtual reality environments, and assistive devices such as hand orthoses and functional electrical stimulators using neural activity recorded with the ECoG sensor.

ELIGIBILITY:
Inclusion Criteria:

* Limited or no ability to use both hands due to cervical spinal cord injury, brachial plexus injury, brainstem stroke, muscular dystrophy, or amyotrophic lateral sclerosis (ALS) or other motor neuron diseases
* At least 1 year post-injury
* Live within 1 hour of the University of Pittsburgh or willing to stay in Pittsburgh while the ECoG electrode is implanted (up to 29 days)
* Additional inclusion criteria must also be reviewed

Exclusion Criteria:

* Certain implanted devices
* Presence of other serious disease or disorder that could affect ability to participate in this study
* Additional exclusion criteria must also be reviewed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Collinger, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Study sponsors, as well as the FDA, will have access to research data and documents in order to monitor the integrity of the study.

REFERENCES:
- [Derived] Degenhart AD, Hiremath SV, Yang Y, Foldes S, Collinger JL, Boninger M, Tyler-Kabara EC, Wang W. Remapping cortical modulation for electrocorticographic brain-computer interfaces: a somatotopy-based approach in individuals with upper-limb paralysis. J Neural Eng. 2018 Apr;15(2):026021. doi: 10.1088/1741-2552/aa9bfb. PMID 29160240
- See also: Brain Computer Interface Research at University of Pittsburgh Medical Center (UPMC) / University of Pittsburgh — http://www.upmc.com/bci

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment included interfacing with local research registry participants, clinical SCI physicians, MDS and ALS groups, and attending conferences attended by eligibility populations
Pre-assignment Details: This study did not include "arms" or group assignments.
Period: Overall Study
Arm/Group | Direct Brain Interface Users
Started | 6
First (1st Implanted) Subject Enrolled | 1 (2011: Individual with cervical spinal cord injury enrolled and was eligible. Implanted in 2011.)
Second Subject Enrolled | 1 (2012: Second participant enrolled. Ineligible.)
Third Subject Enrolled | 1 (2013: Third participant enrolled. Withdrew due to family commitments.)
Fourth Subject Enrolled | 1 (2013: Fourth participant enrolled. Ineligible.)
Fifth (2nd Implanted) Subject Enrolled | 1 (2013: Individual with ALS enrolled and was eligible. Implanted in 2014.)
Sixth (3rd Implanted) Subject | 1 (2014: Individual with brachial plexus injury enrolled and was eligible. Implanted in 2015.)
Completed | 3 (2015: Third implanted subject completed the study. This fulfilled the requirements of our grant.)
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Determined ineligible during screening. | 2

BASELINE CHARACTERISTICS:
Population: All individuals were English speaking, with a disability of at least one hand/arm, but no other health issues which would interfere with or be made worse by study participation.
Arm/Group | Direct Brain Interface Users
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 39 [20 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Able to Successfully Control of a Variety of External Devices Using Neural Data Recorded With ECoG
Description: Participants will attempt to control devices such as computer cursors, virtual reality environments and assistive devices such as hand orthoses or surface functional electrical stimulators using their brain activity recorded through ECoG.
Time Frame: Up to 29 days of device implantation
Population: Individuals with limited or no ability to use one or both hands due to cervical spinal cord injury, brachial plexus injury, brainstem stroke, muscular dystrophy, cerebral palsy or amyotrophic lateral sclerosis (ALS) or other motor neuron disease.
Measure: Number; unit: participants
Arm/Group | Direct Brain Interface Users
Number analyzed (Participants) | 3
participants | 3

2. Secondary Outcome: Number of Participants Able to Achieve Direct Brain Control of Assistive Devices Using an Electrocorticography (ECoG)-Based Brain-computer Interface System
Description: Participants will be asked to perform, attempt, or imagine performing motor tasks while their brain activity is recorded in order to observe the changes in neural activity during each task.
Time Frame: Up to 29 days of device implantation
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Direct Brain Interface Users
Number analyzed (Participants) | 3
participants | 3

ADVERSE EVENTS:
Time Frame: 6 months
Description: The period of enrollment for participants who completed the study approximately 6 months. This included up to 3 months of screening visits, 1 month of testing during implantation, and up to 2 months of follow-up.
Arm/Group | Direct Brain Interface Users
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Direct Brain Interface Users (N=6)
Neck pain following implant surgery (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant's neck was sore for a few days following implant surgery. This type of pain as described in the consent form. Pain subsided after a few days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No